CLINICAL TRIAL: NCT02196025
Title: An Open Label Trial of Sequential Bifrontal Low Frequency Repetitive Transcranial Magnetic Stimulation (r-TMS) in the Treatment of Primary Insomnia
Brief Title: Transcranial Magnetic Stimulation for Treatment of Insomnia
Acronym: TMSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201400335
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Insomnia
Keywords: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Transcranial magnetic stimulation (Experimental): Patients will receive sequential bilateral bifrontal low frequency TMS stimulation daily on weekdays for three weeks. In addition, a Pittsburgh Sleep Quality Index (PSQI), Insomnia severity rating index, Montgomery Asberg Depression Rating Scale, and a sleep diary will be kept.
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — Patients will receive sequential bilateral bifrontal low frequency TMS stimulation daily on weekdays for three weeks. In addition, a Pittsburgh Sleep Quality Index (PSQI), Insomnia severity rating index, Montgomery Asberg Depression Rating Scale, and a sleep diary will be kept.
  Other Names: repetitive Transcranial magnetic stimulation; r-TMS; TMS

SUMMARY:
Transcranial magnetic stimulation (TMS) is a non-invasive brain stimulation technique that has been approved as a treatment of depression in patients that have not responded to a trial of one antidepressant medication. The investigators hypothesize that low frequency TMS exerts inhibitory effect on hyper excitable cortical state in patients with chronic insomnia and therefore is therapeutic. The investigators want to compare the change in insomnia scores between baseline and end of treatment in an open label trial with bifrontal low frequency TMS stimulation in 20 patients with primary insomnia using daily stimulation of 3 weeks (15 week days).

DETAILED DESCRIPTION:
Insomnia is a common clinical problem that affects about 25 million people in the US. Insomnia exacts health and economic consequences well beyond inadequate and non-restorative sleep. It increases healthcare costs, causes or adds to medical and psychiatric comorbidities, cognitive impairments, accidents, absenteeism and reduced quality of life. Treatment of insomnia is difficult and usually needs a multimodal approach incorporating various cognitive and behavioral approaches in addition to medication treatment. TMS and other neurophysiological studies have shown presence of a diffuse cortical hyper-arousal in patients with chronic insomnia. High frequency TMS (>1 Hz) has been shown to be activating whereas low frequency TMS (<1Hz) has been shown to be inhibitory in clinical and neurophysiological studies. TMS has been approved as a treatment of depression in patients who have not responded to a trial of at least one antidepressant medication. The goal of this study is to translate the knowledge learned from neurophysiological studies of insomnia to the clinical treatment of insomnia using TMS as the primary modality.

Aim: Compare the change in insomnia scores between baseline and end of treatment with bifrontal low frequency TMS stimulation in 20 patients with primary insomnia using daily stimulation of 3 weeks (15 week days).

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred for evaluation and management of insomnia to our sleep disorders clinic will be offered enrollment in this study
2. Patients must meet Diagnostic and Statistical Manual (DSM) IV criteria for Primary insomnia
3. Aged 21-65 years to target relatively healthy adults

Exclusion Criteria:

1. Patients with co-morbid depression
2. Substance abuse in last two weeks
3. No Psychotropic medication changes 2 weeks before start of TMS treatment and no changes during the 3 week treatment period
4. Patients with a major medical or psychiatric disorder that may be causing or contributing to insomnia: bipolar disorder, psychosis, anxiety disorders, dementia, seizure disorder and chronic pain
5. Patients with ferromagnetic material in their head or within 30 cm of the coil will be excluded

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Holbert, MD, Principal Investigator — University of Florida
Locations (1):
- UF @ Shands, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were only included in the study if they met all of the inclusion and no exclusion criteria. Participants must have had a primary diagnosis of insomnia in order to qualify.
Groups:
- Transcranial Magnetic Stimulation: Patients will receive sequential bilateral bifrontal low frequency Transcranial Magnetic Stimulation (TMS) daily on weekdays for three weeks. In addition, a Pittsburgh Sleep Quality Index (PSQI), Insomnia severity rating index, Montgomery Asberg Depression Rating Scale, and a sleep diary will be kept.
  Transcranial magnetic stimulation: Patients will receive sequential bilateral bifrontal low frequency TMS stimulation daily on weekdays for three weeks. In addition, a Pittsburgh Sleep Quality Index (PSQI), Insomnia severity rating index, Montgomery Asberg Depression Rating Scale, and a sleep diary will be kept.
Period: Overall Study
Arm/Group | Transcranial Magnetic Stimulation
Started | 23
Completed | 19
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: 19 people were analyzed for the baseline measure
Arm/Group | Transcranial Magnetic Stimulation
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 12
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Pittsburgh Sleep Quality Index ( PSQI)
Description: Change in Pittsburgh sleep quality index scores at the end of three weeks of stimulation with transcranial magnetic stimulation. Minimum Score = 0 (good sleep); Maximum Score = 30 (disrupted sleep)
Time Frame: three weeks
Population: All participants who completed the PSQI at baseline through week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Magnetic Stimulation
Number analyzed (Participants) | 20
score on a scale
  Baseline score | 12.50 (2.74)
  End of week 1 | 11.70 (3.73)
  End of week 2 | 10.37 (4.04)
  End of week 3 | 9.50 (4.27)

2. Secondary Outcome: Insomnia Severity Index ( ISI)
Description: Change in insomnia severity index scores at the end of three weeks stimulation with transcranial magnetic stimulation. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Time Frame: three weeks
Population: All participants who completed the ISI from baseline to week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Magnetic Stimulation
Number analyzed (Participants) | 20
score on a scale
  Baseline | 20.05 (5.14)
  End of week 1 | 18.37 (5.49)
  End of week 2 | 13.94 (7.10)
  End of week 3 | 10.29 (7.74)

ADVERSE EVENTS:
Time Frame: Adverse event data was captured from enrollment through the end of week 3 for each participant
Description: All adverse events (AE) are captured per CT.gov and University of Florida (UF) requirements. AE's are assessed at each visit.
Arm/Group | Transcranial Magnetic Stimulation
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 2/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcranial Magnetic Stimulation (N=23)
Slight right eye twinge (Eye disorders) | 1 (1) — Resolved
Headache (Nervous system disorders) | 1 — Resolved
Pain at stimulation sight (Skin and subcutaneous tissue disorders) | 1 — Resolved

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT02196025/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT02196025/ICF_001.pdf